CLINICAL TRIAL: NCT03581877
Title: Peripheral Low Dose Systemic Thrombolysis Versus Catheter Directed Acoustic Pulse Thrombolysis for Treatment of Submassive Pulmonary Embolism
Brief Title: Peripheral Systemic Thrombolysis Versus Catheter Directed Thrombolysis for Submassive PE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Azhar Supariwala MD, FACC, FASE, Director of Structural Imaging Southside Hospital Northwell Health, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0805
Record Dates: First submitted 2018-05-07; First posted 2018-07-10 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Embolism; Pulmonary Hypertension; Thromboembolism; Right Ventricular Dysfunction
Keywords: Alteplase; submassive pulmonary embolism; Thrombolysis; pulmonary catheter
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary; Thromboembolism; Ventricular Dysfunction, Right | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: This study will be a prospective randomized interventional study. Patients referred to Southside hospital will be consented to take part in the study. After obtaining written informed consent, investigators will subsequently enroll 158 consecutive patients (aged> 18 years) randomized in a serial 1:1 allocation for either low dose PLST or ACDT for submassive pulmonary embolism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Peripheral low dose thrombolysis (Experimental): Peripheral low dose thrombolysis will use a peripheral vein into an arm as in routine intravenous therapy. This is the experimental arm. Alteplate (R-tpa) belong to thrombolytic or fibrnolytic drug class. Routine hospital policies for peripheral venous therapy will be used. A fixed dose of 24 mg of Activase (Atleplase) over 12 hours or 2.0 mg/hr will be administered peripherally. Simultaneously, intravenous unfractionated heparin will be given with a target partial thromboplastin time of 40 to 60 secs.
  Interventions: Drug: Alteplase
- Catheter directed acoustic thrombolysis (Active Comparator): For ACDT, routine hospital protocols and EKOS(generic) will be used. EKOS is made up of 3 parts which include the drug delivery pulmonary artery catheter, a removable microsonic device, and a reusable Eko-Sonic control unit. Venous access will be obtained by ultrasound guidance in the internal jugular vein or femoral vein. After catheter placement, the right heart pressures will be measured. R-tpa will be directly given into the pulmonary catheter. A fixed dose of 24 mg of tpa over 12 hours or 2.0mg/hr will be given. For unilateral PE, a single catheter will be used with infusion rate of 2 mg//hr and two catheters will be used for bilateral PEs each with 1 mg /hr infusion rate. Intravenous unfractionated heparin will be given with a target partial thromboplastin time of 40 to 60 secs.
  Interventions: Device: EKOS

INTERVENTIONS:
Drug: Alteplase — As stated before, low dose r-tpa will be administered through a peripheral vein for PLST.
  Other Names: Peripheral low dose systemic thrombolysis (PLST)
  Arms: Peripheral low dose thrombolysis
Device: EKOS — As stated before, the EKos device will be used for ultrasound assisted catheter directed thrombolysis or ACDT, same dose t-tpa will administered through the pulmonary catheter. It will be given at a fixed dose over 24 hours.
  Other Names: Ultrasound assisted catheter directed thrombolysis (ACDT)
  Arms: Catheter directed acoustic thrombolysis

SUMMARY:
To determine whether peripheral low dose systemic thrombolysis (PLST) is non-inferior to catheter directed acoustic pulse thrombolysis (ACDT) in improving RV function and reducing pulmonary artery pressures in submassive pulmonary embolism (PE)

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) is a life-threatening event associated with high morbidity and mortality. With more than 100,000 deaths per year, PE constitutes the third most common cardiovascular cause of death following myocardial infarction and stroke. In non massive PE, anticoagulation is the treatment of choice. Advanced treatment options such as systemic thrombolysis in submassive and massive PE help reduce mortality but unfortunately are associated with bleeding complications such as a 2 to 5% risk of hemorrhagic stroke.This has led to development of pharmaco-mechanical therapies such as catheter directed thrombolysis (CDT).

Current guidelines advocate against the use of full dose systemic thrombolysis for acute submassive PE in all patients unless the bleeding risk is very low. CDT has shown efficiency in reducing right ventricular strain and pulmonary hypertension without increasing bleeding complications in trial populations. Ultrasound assisted CDT (ACDT) is an established treatment modality for acute PE which utilizes high frequency low power ultrasonic waves. It is FDA approved for sub-massive and massive pulmonary embolism. However, ultrasound does not breakdown the thrombus itself but increases the permeability for thrombolytic drugs. The ULTIMA trial showed ACDT was superior to anticoagulation treatment in reducing pulmonary hypertension (PH) and right ventricular dilatation in submassive and massive PE. The trial also reported no intracranial hemorrhage. The exact benefit and mechanism of ACDT in dissolving clots is still not clear. Recently, the PERFECT registry described 100 patients who underwent CDT (64%) and ACDT (46%) for PE, the study showed no difference in reduction of pulmonary artery pressures.

ACDT requires the placement of catheters in the pulmonary arteries in a catheterization laboratory by an interventional cardiologist/radiologist through the internal jugular vein/femoral vein and catheters are kept for 12-24 hrs to infuse recombinant tissue plasminogen activator (r-tpa). While many healthcare systems have developed a pulmonary embolism response team (PERT) to make a prompt therapeutic decision in submassive and massive pulmonary embolism management. However, it is not uncommon for CDT to be delayed (sometimes > 12 hours) after the initial diagnosis due to the availability of the interventional cardiologist. Furthermore, placement of pulmonary catheters in CDT can have the risk, albeit low, of pulmonary vasculature injury.

The investigators hypothesize that low dose thrombolytic therapy can be administered through a peripheral vein. PLST is rapidly administrable and does not require placement in a catheterization laboratory by an interventional cardiologist. In addition, the use of low dose r-tpa reduces risk of major bleeding complications. The investigators aim to see if equivalent low dose r-tpa given peripherally i.e PLST is non-inferior to ACDT for the treatment of submassive PE. Both treatments will be compared in safety, efficacy and overall cardiopulmonary function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, able to consent
2. Submassive PE evidenced by CT showing saddle pulmonary embolism, central right and/or left main pulmonary artery emboli.
3. Submassive PE confirmed by right ventricular dimension to left ventricular dimension ratio ≥ 1 in apical 4-chamber view echo/CT scan.
4. Signs of RV dysfunction by echocardiogram, or elevated troponin I >0.04, or pro-BNP > 400 on serial measurements.
5. PE symptom duration less than or equal to 14 days -

Exclusion Criteria:

1. Age <18 to age >90 years;
2. PE symptom duration >14 days;
3. Administration of thrombolytic drugs in the last 4 days
4. Contraindications to thrombolytic therapy:

   1. Active bleeding disorder or coagulation disorder;
   2. Platelet count <100 000/mm3
   3. Hematocrit < 30%
   4. INR> 3
   5. Previous history of vitamin K antagonists with international normalized ratio >2.5 on admission
   6. History of intracranial or intraspinal surgery or trauma or intracranial/intraspinal bleeding
   7. Intracranial neoplasm
   8. Arteriovenous malformation, or aneurysm
   9. Gastrointestinal bleeding <3 months
   10. Internal eye surgery or hemorrhagic retinopathy less than three-month duration
   11. Major surgery, cataract surgery, obstetric delivery, cardiopulmonary resuscitation, or invasive procedure less than10 days duration
   12. Allergy, hypersensitivity, or thrombocytopenia caused heparin or tPA
5. Severe contrast allergy to iodinated contrast
6. Large (>10 mm) right atrial or right ventricular thrombus
7. Systolic blood pressure <90 mm Hg
8. Severe hypertension on repeat measurement (systolic >180 mm Hg or diastolic >105 mm Hg)
9. Pregnancy
10. In any other investigational drug or device study
11. Inability to follow instructions or comply with treatment

    -

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2025-03-19 (Estimated)

PRIMARY OUTCOMES:
Right ventricle (RV) to Left ventricle (LV) ratio | 48 hours
  Investigators will measure and compare the change between baseline and 48 hours right ventricular diameter to left ventricular diameter (RV:LV ratio) on echocardiogram after PLST or ACDT
Pulmonary pressures | 48 hours
  Investigators will measure and compare the change between baseline and 48 hours pulmonary pressures (mm Hg) with echocardiogram following therapy with PLST or ACDT therapy.

SECONDARY OUTCOMES:
Mortality | 30 days
  Composite of all-cause mortality and fatal bleeding in-hospital and at 30-day

OTHER OUTCOMES:
Right ventricle (RV) to Left ventricle (LV) ratio | 30 days
  Investigators will measure and compare the change between baseline and 30 days right ventricular diameter to left ventricular diameter (RV:LV ratio) on echocardiogram after PLST or ACDT
Pulmonary pressures | 30 days
  Investigators will measure and compare the change between baseline and 30 days pulmonary pressures (mm Hg) with echocardiogram following therapy with PLST or ACDT therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Azhar Supariwala, MD, Principal Investigator — Southside Northwell Hospital
Locations (2):
- United States (2):
  - Southside Northwell Hospital, Bay Shore, New York
  - Long Island Jewish Medical Center, Queens, New York

IPD SHARING:
Plan to Share IPD: No
Investigators are not planning to share information or participant data with other researchers

REFERENCES:
- [Background] Anderson FA Jr, Wheeler HB, Goldberg RJ, Hosmer DW, Patwardhan NA, Jovanovic B, Forcier A, Dalen JE. A population-based perspective of the hospital incidence and case-fatality rates of deep vein thrombosis and pulmonary embolism. The Worcester DVT Study. Arch Intern Med. 1991 May;151(5):933-8. PMID 2025141
- [Background] Chatterjee S, Chakraborty A, Weinberg I, Kadakia M, Wilensky RL, Sardar P, Kumbhani DJ, Mukherjee D, Jaff MR, Giri J. Thrombolysis for pulmonary embolism and risk of all-cause mortality, major bleeding, and intracranial hemorrhage: a meta-analysis. JAMA. 2014 Jun 18;311(23):2414-21. doi: 10.1001/jama.2014.5990. PMID 24938564
- [Background] Kuo WT, Gould MK, Louie JD, Rosenberg JK, Sze DY, Hofmann LV. Catheter-directed therapy for the treatment of massive pulmonary embolism: systematic review and meta-analysis of modern techniques. J Vasc Interv Radiol. 2009 Nov;20(11):1431-40. doi: 10.1016/j.jvir.2009.08.002. PMID 19875060
- [Background] Jaff MR, McMurtry MS, Archer SL, Cushman M, Goldenberg N, Goldhaber SZ, Jenkins JS, Kline JA, Michaels AD, Thistlethwaite P, Vedantham S, White RJ, Zierler BK; American Heart Association Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; American Heart Association Council on Peripheral Vascular Disease; American Heart Association Council on Arteriosclerosis, Thrombosis and Vascular Biology. Management of massive and submassive pulmonary embolism, iliofemoral deep vein thrombosis, and chronic thromboembolic pulmonary hypertension: a scientific statement from the American Heart Association. Circulation. 2011 Apr 26;123(16):1788-830. doi: 10.1161/CIR.0b013e318214914f. Epub 2011 Mar 21. PMID 21422387
- [Background] Kucher N, Boekstegers P, Muller OJ, Kupatt C, Beyer-Westendorf J, Heitzer T, Tebbe U, Horstkotte J, Muller R, Blessing E, Greif M, Lange P, Hoffmann RT, Werth S, Barmeyer A, Hartel D, Grunwald H, Empen K, Baumgartner I. Randomized, controlled trial of ultrasound-assisted catheter-directed thrombolysis for acute intermediate-risk pulmonary embolism. Circulation. 2014 Jan 28;129(4):479-86. doi: 10.1161/CIRCULATIONAHA.113.005544. Epub 2013 Nov 13. PMID 24226805
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Braaten JV, Goss RA, Francis CW. Ultrasound reversibly disaggregates fibrin fibers. Thromb Haemost. 1997 Sep;78(3):1063-8. PMID 9308755
- [Background] Engelberger RP, Spirk D, Willenberg T, Alatri A, Do DD, Baumgartner I, Kucher N. Ultrasound-assisted versus conventional catheter-directed thrombolysis for acute iliofemoral deep vein thrombosis. Circ Cardiovasc Interv. 2015 Jan;8(1):e002027. doi: 10.1161/CIRCINTERVENTIONS.114.002027. PMID 25593121
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Becattini C, Agnelli G, Salvi A, Grifoni S, Pancaldi LG, Enea I, Balsemin F, Campanini M, Ghirarduzzi A, Casazza F; TIPES Study Group. Bolus tenecteplase for right ventricle dysfunction in hemodynamically stable patients with pulmonary embolism. Thromb Res. 2010 Mar;125(3):e82-6. doi: 10.1016/j.thromres.2009.09.017. Epub 2009 Oct 14. PMID 19833379